CLINICAL TRIAL: NCT00637780
Title: An Open Label Non-randomized Study To Characterize The Steady State Pharmacokinetics Of Sulfasalazine Delayed Release Tablets In Children With Juvenile Idiopathic Arthritis
Brief Title: Study To Determine The Pharmacokinetics Of Sulfasalazine In Children With Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated on 13 April 2016 for business reasons. No safety and/or efficacy concerns contributed to the termination of the study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0031005
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Sulfasalazine delayed release tablets; azulfidine entabs; Pharmacokinetics; Juvenile Idiopathic Arthritis (JIA)
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Sulfasalazine; Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sulfasalazine delayed release tablets 30-60 mg/kg/day (divided into BID doses) for 6 days
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine delayed release tablets 30-60 mg/kg/day (divided into BID doses) for 7 days. Blood sampling for Pharmacokinetic assessment to be performed on Day 7
  Other Names: AZULFIDINE EN-tabs Tablets

SUMMARY:
This study will characterize the steady state pharmacokinetics of sulfasalazine delayed release tablets in pediatric Juvenile Idiopathic Arthritis patients. Data from this study will fulfill the post approval commitment to the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of oligoarticular, polyarticular, psoriatic or enthesitis-related JIA as determined by ILAR criteria. Patients who have been continuously treated with generic sulfasalazine delayed release formulation and have tolerated the product for at least 3 months prior to study enrolment and who are switched to Azulfidine-EN at least 8 days prior to Day 0 are eligible.
* Patients must be at least 6 years of age and has not reached his/her 18th birthday prior to the Baseline Visit (Day 0).
* Onset of JIA must have occurred prior to the patient's 16th birthday.
* Patients must weigh at least 20 kg.
* Patients must be on sulfasalazine 500 mg delayed release tablets and the total daily dose must be within the specified range of 30-60 mg/kg/day with a maximum daily dose of 3 g/day

Exclusion Criteria:

* Patient currently with systemic features of systemic JIA.
* Hypersensitivity to sulfasalazine , its metabolites, sulfonamides or salicylates.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Inability to swallow whole (uncrushed) sulfasalazine 500 mg delayed release tablets as required by protocol

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States
- Private Office, Guadalajara, Jalisco, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0031005&StudyName=Study%20To%20Determine%20The%20Pharmacokinetics%20Of%20Sulfasalazine%20In%20Children%20With%20Juvenile%20Idiopathic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The last participant enrolled in 2014 but the study was kept open for another 2 years and enrollment was not stopped. However, by 2016, no additional participants were enrolled and thus the study was closed. As such, the basic results for this study are only prepared in 2016 though last participant's last visit was in 2014.
Groups:
- Sulfasalazine in Juvenile Idiopathic Arthritis: All participants received sulfasalazine 30-50 milligrams (mg)/kilograms (kg)/day, divided into twice daily (BID) doses, for 6 days. On Day 7, the morning dose was administered at the site in presence of site staff. Sulfasalazine was administered orally in the form of 500-mg tablets.
Period: Overall Study
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The only 2 participants who were enrolled and completed the study at study termination were included in all analyses.
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.4)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Sulfasalazine Steady State Maximum Plasma Concentration (Cmax) and Predose Concentration (Cmin)
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: The 2 participants who were enrolled and completed the study at the time of study termination were included in all analyses.
Measure: Number; unit: micrograms (mcg)/milliliter (mL)
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
micrograms (mcg)/milliliter (mL)
  Cmax - Value 1 | 17.6 [4.51 to 17.6]
  Cmax - Value 2 | 4.51 [0.988 to 4.28]
  Cmin - Value 1 | 4.28
  Cmin - Value 2 | 0.988

2. Primary Outcome: Sulfasalazine Time for Cmax (Tmax) at Steady State
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: hours (hr)
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
hours (hr)
  Value 1 | 2.02
  Value 2 | 5.92

3. Primary Outcome: Sulfasalazine Area Under the Concentration-time Profile From Time 0 to Time Tau, the Dosing Interval (AUCtau) at Steady State
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: mcg*hr/mL
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
mcg*hr/mL
  Value 1 | 110
  Value 2 | 34.7

4. Primary Outcome: Sulfapyridine Steady State Cmax and Cmin
Description: Sulfapyridine and 5-aminosalicylic acid (5-ASA) are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: mcg/mL
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
mcg/mL
  Cmax - Value 1 | 21.7
  Cmax - Value 2 | 7.68
  Cmin - Value 1 | 14.7
  Cmin - Value 2 | 4.79

5. Primary Outcome: Sulfapyridine Tmax at Steady State
Description: Sulfapyridine and 5-ASA are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: hr
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
hr
  Value 1 | 4.00
  Value 2 | 11.9

6. Primary Outcome: Sulfapyridine AUCtau at Steady State
Description: Sulfapyridine and 5-ASA are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: mcg*hr/mL
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
mcg*hr/mL
  Value 1 | 232
  Value 2 | 67.3

7. Primary Outcome: 5-aminosalicylic Acid (5-ASA) Steady State Cmax and Cmin
Description: Sulfapyridine and 5-ASA are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: mcg/mL
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
mcg/mL
  Cmax - Value 1 | 0.208
  Cmax - Value 2 | 0.0982
  Cmin - Value 1 | 0.0439
  Cmin - Value 2 | 0.0816

8. Primary Outcome: 5-aminosalicylic Acid (5-ASA) Tmax at Steady State
Description: Sulfapyridine and 5-ASA are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: hr
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
hr
  Value 1 | 0.000
  Value 2 | 11.9

9. Primary Outcome: 5-aminosalicylic Acid (5-ASA) AUCtau at Steady State
Description: Sulfapyridine and 5-ASA are primary metabolites of sulfasalazine, the study drug.
Time Frame: Day 7 predose, and 2, 4, 6, 10, and 12 hours postdose
Population: as for outcome 1
Measure: Number; unit: mcg*hr/mL
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
mcg*hr/mL
  Value 1 | 1.63
  Value 2 | 1.04

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Withdrawals Due to TEAEs
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAEs are defined as newly occurring AEs or those worsening after first dose. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Screening through to and including 28 calendar days after the last administration of the investigational product
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
participants
  TEAEs | 0
  SAEs | 0
  Withdrawals due to TEAEs | 0

11. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes,clinical chemistry, and urinalysis (dipstick and microscopy).
Time Frame: Screening, Day 0, and Day 7
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
participants | 1

12. Secondary Outcome: Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria
Description: Vital sign values which met categorical summarization criteria included: supine/sitting pulse rate less than (<) 40 or more than (>) 120 beats per minute (bpm); erect pulse rate <40 or >140 bpm; changes from baseline in same posture of systolic blood pressure (SBP) more than or equal to (>=) 30 millimeters of mercury (mm Hg) or diastolic blood pressure (DBP) >=20 mm Hg; SBP <90 mm Hg; and DBP <50 mm Hg.
Time Frame: Screening, Day 0, and Day 7
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: Screening through to and including 28 calendar days after the last administration of the investigational product.
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sulfasalazine in Juvenile Idiopathic Arthritis
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated prematurely and only 2 participants were enrolled and completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.